CLINICAL TRIAL: NCT06737588
Title: The Addictive Diagnostic Value of Apparent Diffusion Coefficients to PI-RADS 3-5 of Biparametric Magnetic Resonance Imaging in the Diagnosis of Prostate Cancer
Brief Title: The Addictive Diagnostic Value of Apparent Diffusion Coefficients to bpMRI in the Diagnosis of Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, XiaoJun, Professor, Chief Physician, Anhui Provincial Hospital
Other Study IDs: 2024-ky-495 (bpMRI-ADC)
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Prostate biospy; Biparametric Magnetic Resonance; Apparent diffussion coefficient; Prostate Imaging-Reporting and Data System; Diagnosis
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to evaluate the diagnostic value of different ADC values (incuding ADCmin, ADCmean, ADCratio and ADCrange) of bpMRI in patients with PI-RADS 3-5. The main aim is to evaluate whether different ADC values improve the diagnosis of clinically significant prostate cancer (Gleasonscore≥3+4, ISUP grade ≥2) and any-grade prostate cancer (Gleasonscore≥3+3, ISUP grade ≥1).

DETAILED DESCRIPTION:
The study is conducted with suspected prostate cancer. Patients with PI-RADS scores of 3-5 after completing prostate bpMRI chose to undergo prostate biopsy. Before patients undergo prostate biopsy, researchers will collecte information on age, BMI, tPSA, f/PSA, PV, PSAD, ADCmean, ADCmin, ADCmax, ADCnormal, maximum lesion diameter, location of major lesions, and so on. For prostate biopsy, systematic prostate biopsy ± bpMRI cognitive fusion targeted prostate biopsy will be completed under the conditions permitted by physical condition, and Gleason score will be clearly given by pathologists if the final diagnosis is prostate cancer. In this study, the pathological result is regarded as the gold standard. ROC curve, area under curve, sensitivity, specificity, positive predictive value, negative predictive value, positive likelihood ratio, negative likelihood ratio and other indicators of diagnostic test were calculated. Relevant conclusions are finally drawn by comparing the diagnostic capacity of different ADC values for prostate cancer. Meanwhile, binary logistic regression analysis will also conduct the Odds ratios (ORs) and 95% confidence intervals (CIs) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. The patient met at least one indication of prostate biopsy (Chinese expert consensus on prostate biopsy (2022 edition) https://rs.yiigle.com/cmaid/1442948 );
2. Serum PSA test was completed in the patient with tPSA < 100 ng/ml;
3. Primary prostate tumor lesion, no history of other tumors;
4. Completed 3.0T bpMRI examination, PI-RADS score ≥3 score, the image is clear and readable;
5. Patients fully understand the relevant contents of the study and voluntarily sign the informed consent.

Exclusion Criteria:

1. The patient has contraindications for MRI;
2. PI-RADS 1-2 of bpMRI;
3. The patient had contraindications to prostate biopsy or explicitly refused biopsy;
4. bpMRI indicated that the patient had multiple lymph nodes or bone metastases;
5. Previous prostate-related surgery;
6. The patient refused to sign the informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is observational and does not require any intervention for patients, who only need to complete the routine diagnosis and treatment procedures. This study mainly screened patients who need to complete mainly included serum PSA test, digital rectal examination, and 3.0TbpMRI containing ADC maps and with indications of prostate biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate whether ADC values can improve the diagnostic capacity of bpMRI for clinically significant prostate cancer (csPCa) (Gleason score ≥ 3+4, ISUP grade ≥ 2) in patients with PI-RADS 3-5. | through study completion, an average of 1 month
  csPCa means Gleason score ≥ 3+4， ISUP grade ≥ 2. Evaluation indexes: ROC curves and AUC value (95%CI) , Sensetivity, Specificity, Positive predictive value and negative predictive value. The odds ratios (ORs) and 95% confidence intervals in logistic analysis.

SECONDARY OUTCOMES:
Evaluate whether ADC values can improve the diagnostic capacity of bpMRI for any-grade prostate cancer (PCa) (Gleason score ≥ 3+3, ISUP grade ≥ 1) in patients with PI-RADS 3-5. | through study completion, an average of 1 month
  agPCa means Gleason score ≥ 3+3， ISUP grade ≥ 1. Evaluation indexes: ROC curves and AUC value (95%CI) , Sensetivity, Specificity, Positive predictive value and negative predictive value. The odds ratios (ORs) and 95% confidence intervals in logistic analysis.
Evaluate the diagnostic capacity of different PI-RADS scores combined with different ADC cut off values for csPCa | through study completion, an average of 1 month
  ROC curves and AUC value (95%CI), Sensetivity, Specificity, Positive predictive value and negative predictive value.
Compare the diagnostic value of different ADC values for csPCa in patients with 3-5 points of PI-RADS. | through study completion, an average of 1 month
  ROC curves and AUC value (95%CI), Sensetivity, Specificity, Positive predictive value and negative predictive value.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Xiao, Principal Investigator — The First Affiliated Hospital of USTC
Locations (2):
- China (2):
  - Department of Urology, The First Affiliated Hospital of USTC, Division of Life Sciences and Medicine, University of Science and Technology of China, Hefei, Anhui
  - Department of Urology, The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui

IPD SHARING:
Plan to Share IPD: Undecided